CLINICAL TRIAL: NCT00886119
Title: Lotrafilcon B Multifocal Evaluations - Comparison to a Traditional Multifocal in Higher Spectacle Adds
Brief Title: Comparison of a Multifocal Contact Lens to a Traditional Multifocal Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P-319-C-005 sub 8
Record Dates: First submitted 2009-04-10; First posted 2009-04-22 (Estimated); Results first posted 2010-10-29 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-01

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Lotrafilcon B / Omafilcon A (Other): Lotrafilcon B, followed by Omafilcon A
  Interventions: Device: Lotrafilcon B multifocal contact lens; Device: Omafilcon A multifocal contact lens
- Omafilcon A / Lotrafilcon B (Other): Omafilcon A, followed by Lotrafilcon B
  Interventions: Device: Lotrafilcon B multifocal contact lens; Device: Omafilcon A multifocal contact lens

INTERVENTIONS:
Device: Lotrafilcon B multifocal contact lens — Silicone hydrogel, soft, multifocal contact lens for daily wear use
Device: Omafilcon A multifocal contact lens — Hydrogel, soft, multifocal contact lens for daily wear use

SUMMARY:
The purpose of the trial is to compare the performance of two multifocal contact lens systems/products in established presbyopic subjects.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 35 years of age.
* Best-corrected visual acuity of at least 20/40 in each eye.
* Spectacle add from +1.50D and +2.50D (inclusive).
* Able to be fit in available study sphere powers (Plano to -4.00D).
* Currently wearing soft contact lenses at least 5 days a week.
* Other protocol inclusion / exclusion criteria may apply.

Exclusion Criteria:

* Requires concurrent ocular medication.
* Eye injury or surgery within twelve weeks immediately prior to enrollment.
* Currently enrolled in an ophthalmic clinical trial.
* Evidence of systemic or ocular abnormality, infection or disease likely to affect successful wear of contact lenses or use of their accessory solutions.
* Previous refractive surgery.
* Astigmatism > 1.00D.
* Currently wearing Proclear Multifocal, Frequency 55 Multifocal or Biomedics EP contact lenses.
* Other protocol inclusion / exclusion criteria may apply.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants were enrolled but not dispensed due to failing inclusion/exclusion criteria. These participants were included in the Actual Enrollment calculation, but not Participant Flow or Baseline Characteristics calculations.
Groups:
- Lotrafilcon B / Omafilcon A: Lotrafilcon B multifocal contact lens worn first, with Omafilcon A multifocal contact lens worn second. Both products worn in a daily wear basis.
- Omafilcon A / Lotrafilcon B: Omafilcon A multifocal contact lens worn first, with Lotrafilcon B multifocal contact lens worn second. Both products worn in a daily wear basis.
Period: Period 1
Arm/Group | Lotrafilcon B / Omafilcon A | Omafilcon A / Lotrafilcon B
Started | 24 | 22
Completed | 23 | 22
Not Completed | 1 | 0
Not completed — Did not meet inclusion criteria | 1 | 0
Period: Period 2
Arm/Group | Lotrafilcon B / Omafilcon A | Omafilcon A / Lotrafilcon B
Started | 23 | 22
Completed | 23 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed subjects.
Arm/Group | Overall
Number analyzed (Participants) | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 49.3 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Corrected Distance Binocular Visual Measurement in Normal Illumination Reported as Binocular Distance Visual Acuity
Description: Tested while reading charts distant to the subject with both eyes together in normal lighting. This outcome is measured in logMAR units (logarithm of the minimum angle of resolution). A logMAR acuity of 0.0 equates to 20/20 Snellen acuity and is considered normal. Positive logMAR values indicate poorer vision and negative values denote better visual acuity.
Time Frame: After 1 week of wear
Population: Per Protocol. Analysis excluded major protocol deviations as determined by masked review.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Lotrafilcon B: Silicone hydrogel, soft, multifocal contact lens for daily wear use
- Omafilcon A: Hydrogel, soft, multifocal contact lens for daily wear
Arm/Group | Lotrafilcon B | Omafilcon A
Number analyzed (Participants) | 36 | 41
logMAR | 0.00 (0.07) | -0.02 (0.06)

ADVERSE EVENTS:
Time Frame: 7 weeks, the duration of the trial.
Groups:
- Lotrafilcon B: Silicone hydrogel, soft, multifocal contact lens for daily wear
Arm/Group | Lotrafilcon B | Omafilcon A
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/45
Other Adverse Events (participants affected / at risk) | 0/46 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any pre-clinical and/or clinical data or impressions from this trial.